CLINICAL TRIAL: NCT02971709
Title: Norms and Built Environment: Use of Shade in U.S. and Australian City Parks
Brief Title: Use of Shade in U.S. and Australian City Parks
Acronym: Shade
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klein Buendel, Inc. (Industry)
Collaborators: Cancer Council Victoria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CA140367; 0265 (Other: Klein Buendel, Inc.)
Record Dates: First submitted 2016-11-21; First posted 2016-11-23 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Skin Cancer
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Shade Sail (Experimental): Shade sails were constructed over passive recreation areas in public parks between pretest and posttest. Shade sails maximized available shade in the passive recreation areas from 11 am to 3 pm in the summer.
  Interventions: Behavioral: Shade Sail
- Unshaded Control (No Intervention): Passive recreation areas in public parks that remained unshaded at pretest and posttest.

INTERVENTIONS:
Behavioral: Shade Sail — Shade sails had powder-coated or gout galvanized steel poles and a lighter colored shade cloth to transmit visual light. The shade cloth met Ultraviolet Protection Factor (UPF) ratings to reduce UV under the shade cloth by 94%. The final shade sail designs and sizes were determined with input from parks department staff and complied with all local engineering, building, and planning codes. Shade sails exceeded the minimum safety requirements for strength (for wind and snow load), resistance to light degradation, and UV transmission. The design minimized climbing access points and hazards to adjacent activities.
  Arms: Shade Sail

SUMMARY:
Use of shade when outdoors is recommended by health authorities worldwide to reduce overall exposure to ultraviolet radiation. However, expensive physical environment changes are often required to provide shade and may be effective only when health education has created a social environment that motivate shade use. A multi-national research team will explore the use of built shade in passive recreation areas within public parks and compare use of built shade between the United States and Australia. The specific aims of the project are to: a) introduce built shade structures (i.e., shade sails) in public parks in Denver and Melbourne; b) compare the use of passive recreation areas with and without built shade; c) compare the change in use of the passive recreation areas in Denver and Melbourne after introduction of built shade, and d) examine the relationship among social environment and physical features of the environment and built shade.

DETAILED DESCRIPTION:
This study is designed to understand the value of shade development in skin cancer prevention and test predictions from social ecologic models that health behavior results from the interplay among the built environment, social environment, and setting features. Use of shade is recommended by health authorities worldwide. However, shade provision requires expensive physical environment changes and may be effective only when health education has created a social environment (e.g., norms) that motivates its use. A multi-national research team will explore the use of built shade in passive recreation areas (i.e., areas for sitting/ standing while socializing, preparing/eating a meal, watching/coaching sports, watching a concert, taking a class, or waiting, or areas where people stroll for sightseeing, while observing outdoor displays, or shopping) within public parks and compare use between the United States (i.e., Denver, Colorado) and Australia (i.e., Melbourne, Victoria) to prospectively test the moderating influence of social environment on the built environment. Pilot studies confirmed that adults in Melbourne had stronger sun protection habits and norms than adults in Denver. The specific aims of the project are to: a) introduce built shade structures (i.e., shade sails) in public parks in Denver and Melbourne; b) compare the use of passive recreation areas with and without built shade; c) compare the change in use of the passive recreation areas in Denver and Melbourne after introduction of built shade, and d) examine the relationship among social environment and physical features of the environment and built shade.The research team will build shade sails at passive recreation areas in public parks and compare use of the passive recreation areas to unshaded passive recreation areas in a randomized pretest-posttest controlled design. Passive recreation areas will be enrolled in one of three annual sample waves and stratified by location (72 in Denver and 72 in Melbourne). In each wave, passive recreation areas will be pretested in a first summer, further stratified based on baseline use, and randomized following pretest to construction of a shade sail or an untreated control group in a 1:3 ratio. Posttesting will occur the following summer, after construction of the shade sails. In total, 36 passive recreation areas will be randomized to the intervention group with shade sail construction (18 per city) and 108 passive recreation areas to the untreated control group with no shade sails (54 per city). The primary outcome measure will be use of the passive recreation areas, observed by trained research assistants. The secondary outcome measure will be the potential ultraviolet radiation exposure, assessed by hand-held meters during the observations of the passive recreation areas. Data collection will occur during 30-minute periods between 11 am and 3 pm on on 4 weekend days over 20-weeks in the summer. Primary analyses will be performed on the probability the passive recreation areas are in use when observed and secondary analysis, on estimated standard erythemal dose of ultraviolet radiation during 30 minutes, using intent-to-treat methods.

ELIGIBILITY:
Inclusion Criteria:

* Passive recreation areas had to be located in public parks in Denver, Colorado USA or Melbourne, Victoria Australia metropolitan area.
* Parks had to contain at least two unshaded PRAs and be administered by the study municipalities,
* Passive recreation areas had to meet the definition of a passive recreation area, i.e., areas for sitting/standing while socializing, preparing/eating a meal, watching or coaching sports, watching a concert, taking a class, or waiting, or areas where people stroll (walk slowly) for sightseeing while observing outdoor displays (e.g., festivals, gardens, zoo exhibits).
* Passive recreation areas had to be in full sun (i.e. no shade) at pretest.
* Passive recreation areas had to contain a space where a shade sail could be constructed, i.e., free from underground or above ground obstructions, relatively level, and large enough to accommodate the shade sail.
* Passive recreation areas had to be approved by parks department staff for shade sail construction.
* Adults had to appear to be 18 years of age or older.
* Adults had to be in the public parks.

Exclusion Criteria:

* Passive recreation areas where major construction/ redevelopment of the parks was planned within the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2010-07; Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Observed Use of Passive Recreation Area by Adults | One-year
  Any use of each passive recreation, assessed by observing each passive recreation areas for 30 minutes on four weekend days between 11 am and 3 pm when forecast high temperatures were had forecast high temperature were between 72°F/22°C and 95°F/35°C over a 20-week period during two summers (pretest summer, posttest summer) by trained research assistants. Observations were suspended during rain.

SECONDARY OUTCOMES:
Solar Ultraviolet Radiation Level | One-year
  Average potential UV exposure for a user of the passive recreation area assessed in standard erythemal units, based on measurements from a handheld UV meter performed by trained research assistants during assessment of the primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: David Buller, PhD, Principal Investigator — Klein Buendel, Inc.
Locations (2):
- Klein Buendel, Inc., Golden, Colorado, United States
- Cancer Council Victoria, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Buller DB, English DR, Buller MK, Simmons J, Chamberlain JA, Wakefield M, Dobbinson S. Shade Sails and Passive Recreation in Public Parks of Melbourne and Denver: A Randomized Intervention. Am J Public Health. 2017 Dec;107(12):1869-1875. doi: 10.2105/AJPH.2017.304071. Epub 2017 Oct 19. PMID 29048958